CLINICAL TRIAL: NCT06116422
Title: Nutrition and Obesity in Under-Represented Populations: Food Insecurity Research to Advance Science and Improve Health: A Multi-disciplinary Approach for Study and Mitigation of Food Insecurity and Obesity
Brief Title: Nutrition and Obesity in Under-Represented Populations: Food Insecurity Research to Advance Science and Improve Health
Acronym: NOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00114248
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Obesity; Food Insecurity; Nutrition, Healthy; Nutrition Poor
MeSH Terms: conditions — Pediatric Obesity; Malnutrition

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cash Benefit Group (Active Comparator): Provides financial support weekly, in the form of an unrestricted cash benefit. The investigators will partner with Held to provide the card to participants, load the card with $50/week for the 12 months of enrollment, and view the purchases at the vendor level using an existing dashboard Held maintains. Participants will also receive a monthly nutrition guidance brochure tailored to the infant's developmental stage.
  Interventions: Behavioral: Grocery intervention - unrestricted
- Grocery Benefit Group (Active Comparator): Provides financial support weekly in the form of a grocery benefit. The investigators will enroll participants in the Food Lion MVP program, linking the account to a Duke email address. The study team will work with the participants to order $50 worth of groceries from Food Lion, for the participants to pick up from the store. Groceries will be ordered weekly for the 12 months of enrollment and coordinators will have access to view items purchased at Food Lion by each participant.
  Interventions: Behavioral: Grocery intervention - restricted

INTERVENTIONS:
Behavioral: Grocery intervention - unrestricted — Receives financial support in an unrestricted fashion (i.e., can use the money for whatever they need).
  Arms: Cash Benefit Group
Behavioral: Grocery intervention - restricted — Receives financial support restricted to the purchase of items at a grocery store, and with monthly grocery shopping coaching from a trained nutrition expert.
  Arms: Grocery Benefit Group

SUMMARY:
Food insecurity is associated with obesity in children, and childhood obesity leads to long term health consequences. While existing research shows that food benefit programs reduce food insecurity, little is known about the mediating factors between food benefit programs and child health. The purpose of this study is to understand if the resolution of food insecurity in young children with early onset obesity can improve body mass index (BMI) over one year, and if so, by what mechanisms. The investigators will conduct a randomized comparative effectiveness study among infants (n=228) aged 12 months at risk for food insecurity and deliver two different food security interventions. Both will provide families with $50/week for one year of study enrollment. The first group will receive this as an unrestricted cash benefit ("cash benefit group") and the second group will receive this as a benefit in the form of weekly grocery purchases with the support of a trained nutrition expert to guide healthy grocery purchasing ("grocery benefit group"). The investigators will also construct a contemporary comparison cohort of infants meeting the inclusion/exclusion criteria from the electronic health record, using propensity score matching to allow comparisons between both intervention groups and usual care. The primary endpoint is difference in BMI at 12 months post-enrollment (24 months of age). Secondary outcomes include measures of nutrition, food security, electronic health record data related to general child health, and other factors related to parental stress and unmet social needs. Patients will have the opportunity to participate in post-study interviews to report on intervention satisfaction, and facilitators and barriers of infant feeding. Data analysis will be conducted by a trained statistician (Duke Biostatistics, Epidemiology, and Research Design; BERD) and will employ a two-means test for a repeated-measures design. The benefits to participants outweigh the minimal risks of loss of privacy, and confidential information will be managed carefully to minimize this risk.

ELIGIBILITY:
Inclusion:

* Aged 9-12 months and their primary caregiver "parent".
* Medicaid and WIC-eligible (proxy for "at risk for food insecurity")
* World Health Organization BMI ≥ 85%ile at current or most recent encounter (early-onset obesity) OR ≥ 20 pounds at 9 months old.
* Caregiver speaks either English or Spanish as their primary language.
* Infant was born as a singleton infant.

Exclusion:

* Diagnosed with monogenic obesity.
* Plans to move from the area in the next 12 months.
* Parent is currently pregnant.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 228 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in BMI (Body Mass Index) | 1 year
  At 12 months post-enrollment (24 months of age).

OTHER OUTCOMES:
Change in Food Security | baseline, 3, 6, 9 and 12 months
  As measured by an 18 item food insecurity screen to assess food insecurity levels.
Change in Infant Dietary Quality | baseline, 6 months, and 12 months
  As measured by the USDA multipass food recall tool (ASA24).
Change in Unmet social needs | baseline, 6 months, and 12 months
  Changes in social determinants of health affecting the family as measured by the HealthLeads questionnaire.
Perceived stress scale | baseline, 6 months, and 12 months
  As measured by a 10 item perceived stress scale for parents.

CONTACTS AND LOCATIONS:
Locations (1):
- North Duke Street Pediatrics, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No